CLINICAL TRIAL: NCT06768021
Title: Does a Pre-sedation Guided Visualization Exercise Improve Outcomes in Ambulatory Anesthesia for Oral and Maxillofacial Surgery: a Double-blinded, Randomized Controlled Trial
Brief Title: Does Style of Pre-sedation Instructions Improve Patient Outcomes in Ambulatory Anesthesia for Oral and Maxillofacial Surgery?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alameda Health System (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Omid Akramian, Resident Surgeon, Alameda Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB24-10151A; 24-42546 (Other: University of California, San Francisco)
Record Dates: First submitted 2024-12-31; First posted 2025-01-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia Outcomes; Anesthesia Complication; Anesthesia and Procedure Related Time Intervals; Anesthesia Recovery Period; Anesthesia, Intravenous; Anesthesia Induction
Keywords: Anesthesia Experience Survey; Ambulatory anesthesia; Intravenous sedation; Guided Visualization; Pre-sedation instructions; Anesthesia outcomes; Oral & Maxillofacial Surgery (OMFS); Face, Legs, Activity, Cry, Consolability (FLACC)
MeSH Terms: conditions — Facies; Motor Activity; Crying

STUDY DESIGN:
Intervention Model Description: Member(s) of the research team will reference the subject list and determine whether this subject is in the control or experimental group. Based on this grouping, the research team member will enter the operatory and give the corresponding style of standardized pre-sedation instructions to the subject.
  The control group will receive standardized pre-sedation instructions. The intervention group will receive the same set of standardized pre-sedation instructions and a one-minute guided visualization. Once complete, the research team member(s) will leave the operatory and hand back off to the clinical team.
  The clinical team will then administer the anesthetic and perform the surgery, recording amounts of medication delivered and FLACC scores at three points during the case (during local anesthesia, during the surgery, and 15-minutes after surgery).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized pre-sedation instructions only group (Placebo Comparator): This group will receive the standardized pre-sedation instructions only, with no guided visualization.
  Interventions: Behavioral: Standardized pre-sedation instructions only
- Guided visualization and standardized pre-sedation instructions group (Experimental): This arm will receive standardized pre-sedation instructions, as well as one-minute guided visualization.
  Interventions: Behavioral: Guided visualization and standardized pre-sedation instructions

INTERVENTIONS:
Behavioral: Guided visualization and standardized pre-sedation instructions — One arm will receive standardized pre-sedation instructions, as well as one-minute guided visualization.
  Arms: Guided visualization and standardized pre-sedation instructions group
Behavioral: Standardized pre-sedation instructions only — One arm will receive standardized pre-sedation instructions only.
  Arms: Standardized pre-sedation instructions only group

SUMMARY:
This randomized controlled trial aims to evaluate the impact of a brief guided visualization exercise on anesthesia-related outcomes in oral and maxillofacial surgery in patients scheduled for ambulatory anesthesia in the oral and maxillofacial surgery clinic. Researchers will compare these patients, who will receive the guided visualization exercise in addition to standardized pre-operative instructions, to patients who will only receive the standardized pre-operative instructions. The following outcomes will be measured for both groups:

* A seven-point Anesthesia Experience Survey
* Face-Legs-Activity-Cry-Consolability (FLACC) scores at three points in time during the anesthetic - during local anesthesia, during surgery, and fifteen minutes after surgery has concluded
* Amount of medications used during the sedation
* Length of sedation

ELIGIBILITY:
Inclusion Criteria:

* Subjects within ages 8 to 70.
* Subjects planned for ambulatory intravenous sedation in the oral and maxillofacial surgery clinic.
* Ability to understand verbal English or understand instructions using a sign-language or voice interpreter of their native language.

Exclusion Criteria:

* Subjects who cannot understand the instructions, even with an interpreter (extremes of age, cognitive impairments, severe psychiatric disease that may affect participation)
* Subjects not undergoing intravenous sedation (oral sedation, nitrous oxide, local anesthesia)
* Subjects undergoing anesthesia in other environments (gastrointestinal suite, operating rooms, interventional radiology)

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Anesthesia Experience Survey | Within 2 hours of the completion of surgery
  A seven-point survey given after the patient meets Aldrete score discharge criteria, asking the following: how the patient rates their pre-operative anxiety level (0-10), if the patient has any recall of surgery (0 for none, 1 for a little, 2 for everything), if the patient remembers any pain during surgery (0 for none, 1 for a little, 2 for a lot), if the patient feels any nausea (0 for none, 1 for a little, 2 for a lot, 3 for vomiting), if the patient feels any pain now (0 for none, 1 for a little, 2 for a lot), if the patient feels any itching (0 for none, 1 for a little, 2 for a lot), and how satisfied the patient is overall with the sedation/anesthesia experience (0-10).
Face-Legs-Activity-Cry-Consolability (FLACC) | During local anesthesia, during surgery, and fifteen minutes after surgery has concluded
  Face-Legs-Activity-Cry-Consolability (FLACC) is a behavioral scale primarily designed for scoring postoperative pain in infants and young children, but can also be used to assess intraoperative and postoperative pain in adults undergoing intravenous sedation.
  The scale gives 0, 1, or 2 points for each of the following: the appearance of the patient's face, the appearance of the patient's legs, the amount of activity, the presence of crying, and the extent of consolability, for a total of 10 points. 0-3 points corresponds to mild pain, 4-6 to moderate pain, and 7-10 to severe pain.
  The scores will be taken at three points in time during the anesthetic - during local anesthesia, during surgery, and fifteen minutes after surgery has concluded.
Amount of medications used during the sedation | During the sedation
  The amount of each medication utilized during the sedation will be documented.
Length of sedation | During the sedation
  The length of sedation will be measured, with the start point as the administration of the first sedative medication, and the endpoint as the end of phase I of anesthesia recovery, which will be determined with the Aldrete Scoring System.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral & Maxillofacial Surgery Clinic, Highland Hospital, Alameda Health System, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No